CLINICAL TRIAL: NCT00017641
Title: Phase I Study of Immune Ablation and CD34+ Peripheral Blood Stem Cell Support in Patients With Systemic Lupus Erythematosus
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northwestern Memorial Hospital (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/14976; NU-95LU1
Record Dates: First submitted 2001-06-06; First posted 2001-06-06 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-11

CONDITIONS: Systemic Lupus Erythematosus
Keywords: arthritis & connective tissue diseases; immunologic disorders and infectious disorders; rare disease; systemic lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis; Connective Tissue Diseases; Immune System Diseases; Communicable Diseases; Rare Diseases | interventions — Antilymphocyte Serum; Cyclophosphamide; Filgrastim

INTERVENTIONS:
Drug: anti-thymocyte globulin
Drug: cyclophosphamide
Drug: filgrastim
Procedure: CD34+ Peripheral Blood Stem Cell Reinfusion

SUMMARY:
OBJECTIVES:

I. Determine the safety of immune ablation with high-dose cyclophosphamide and anti-thymocyte globulin followed by peripheral blood stem cell support in patients with systemic lupus erythematosus.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients receive cyclophosphamide IV over 1 hour for 2 doses. Patients receive filgrastim (G-CSF) subcutaneously (SC) beginning 24 hours after completion of cyclophosphamide and continuing until leukapheresis is complete. Leukapheresis continues daily until target number of cells is harvested. CD 34+ cells are isolated from peripheral blood stem cells (PBSC) in vitro.

Patients then receive cyclophosphamide IV over 1 hour on days -5 to -2, anti-thymocyte globulin IV over 10 hours on days -4 to -2, and G-CSF SC beginning on day 0 and continuing until blood counts recover. Patients undergo reinfusion of CD34+ PBSC on day 0.

Patients are followed weekly for 90 days, monthly for 1 year, and at 2 years.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Diagnosis of systemic lupus erythematosus with 1 of the following malignant features:

* Nephritis (WHO class III or IV)
* Failed NIH short-course cyclophosphamide therapy
* Vasculitis/immune complex deposition causing end organ signs or symptoms (e.g., cerebritis, transverse myelitis, pulmonary hemorrhage, cardiac failure, or renal failure)
* Hematologic cytopenias that are immune mediated and uncontrolled by conservative measures with any of the following:

Transfusion-dependent anemia with untransfused hemoglobin less than 8 g/dL

Platelet count less than 40,000/mm3 (without transfusions)

Granulocyte count less than 1,000/mm3

Catastrophic anti-phospholipid syndrome

--Patient Characteristics--

Cardiovascular:

* LVEF at least 35%
* No lupus-induced myocarditis
* No history of unstable angina

Pulmonary:

* FEV1/FVC at least 50% predicted
* DLCO at least 50% predicted

Other:

* HIV negative
* No prior or concurrent malignancy except localized basal cell or squamous cell skin cancer
* No uncontrolled diabetes mellitus
* No medical illness that would preclude study
* No psychiatric illness or mental deficiency that would preclude study
* No known hypersensitivity to E. coli-derived proteins
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

Ages: 0 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10
Dates: Start 2001-04

CONTACTS AND LOCATIONS:
Overall Officials: Ann Traynor, Study Chair — Northwestern Memorial Hospital
Locations (2):
- United States (2):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin